CLINICAL TRIAL: NCT07333079
Title: Evaluation of the Effectiveness of Biofeedback Rehabilitation in People After Stroke
Brief Title: Rehabilitation With Biofeedback for People After Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rzeszow (Other)
Responsible Party: Principal Investigator, Justyna Leszczak, Principal Investigator, University of Rzeszow
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Stroke rehabilitation
Record Dates: First submitted 2025-12-27; First posted 2026-01-12 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Rehabilitation; Stroke
Keywords: Rehabilitation; Late period in stroke; Health-resort based rehabilitation; Conventional (traditional) rehabilitation; Modern technologies; Biofeedback
MeSH Terms: conditions — Stroke | interventions — Equipment and Supplies

STUDY DESIGN:
Intervention Model Description: Random selection into groups (study group I, study group II and control group).
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I-Biofeedback method using the Biometrics E-link device and Health-resort based rehabilitation (Experimental): The rehabilitation program will last three weeks, Monday through Friday. Patients will benefit from group and individual exercises (active and assisted exercises, manipulative exercises, PNF-based exercises, balance and breathing exercises), manual massage, and physical treatments such as laser therapy, jacuzzi, mud packs, carbonic acid therapy, TENS therapy, BIO-V lamp, and local cryotherapy. Additionally, patients will receive 30 minutes per day of hand biofeedback training using the Biometrics E-link device.
  Interventions: Other: Biofeedback method using the Biometrics E-link (group I) and Stella Bio (group II) devices.
- Group II -Biofeedback method using the Stella Bio device and Health-resort based rehabilitation. (Experimental): The rehabilitation program will last three weeks, Monday through Friday. Patients will benefit from group and individual exercises (active and assisted exercises, manipulative exercises, PNF-based exercises, balance and breathing exercises), manual massage, and physical treatments such as laser therapy, jacuzzi, mud packs, carbonic acid therapy, TENS therapy, BIO-V lamp, and local cryotherapy. Additionally, patients will receive 30 minutes per day of hand biofeedback training using the Stella Bio device.
  Interventions: Other: Biofeedback method using the Biometrics E-link (group I) and Stella Bio (group II) devices.
- Health-resort based rehabilitation. (No Intervention): Health-resort based rehabilitation Control group - health-resort based treatments, without biofeedback training.
  Health-resort based rehabilitation The rehabilitation programme will last 3 weeks from Monday to Friday. Patients will receive: group and individual exercises (active and assisted exercises, manipulative exercises, PNF-based exercises, balance and breathing exercises), manual massage, physical treatments such as laser, whirlpool, mud packs, carbonic acid therapy , TENS therapy, BIO-V lamp, local cryotherapy

INTERVENTIONS:
Other: Biofeedback method using the Biometrics E-link (group I) and Stella Bio (group II) devices. — Patients in study groups I and II will also receive 30 minutes daily of hand biofeedback training using the Biometrics E-link device (group I) and hand biofeedback training using the Stella Bio device (group II).
  Arms: Group I-Biofeedback method using the Biometrics E-link device and Health-resort based rehabilitation; Group II -Biofeedback method using the Stella Bio device and Health-resort based rehabilitation.

SUMMARY:
The aim of the research will be to evaluate rehabilitation using the biofeedback method in people after stroke.

DETAILED DESCRIPTION:
Study participants will be randomly assigned to a study group and a control group.

* Study group I - will complete a conventional rehabilitation program supplemented with biofeedback exercises using the Biometrics E-link device
* Study group II - will complete a conventional rehabilitation program supplemented with biofeedback exercises using the Stella Bio device
* Control group - will complete a standard spa rehabilitation program without biofeedback exercises.

The study participants will be patients admitted to the Spa and Rehabilitation Hospital in Iwonicz-Zdrój, Poland, after a late-stage stroke.

Patients will undergo continuous inpatient rehabilitation (3 weeks). The first examination will be conducted on the day of hospital admission, the second on the day of discharge, and the third (follow-up) 3 months after hospital discharge, during a follow-up visit.

Prior to the study, a socio-demographic questionnaire will be administered, including questions about education, marital status, and place of residence.

Measurements will be performed three times for all participants:

* hand muscle strength assessment
* calculated body mass index (BMI)
* proprioceptive testing (mirror test, Thumb Location Test)
* rehabilitation outcome assessment
* functional capacity - Barthel Index, ADL
* Ashworth muscle tone (spasticity)
* hand dexterity using the Box and Blocks test
* hand grip function according to the Frenchay scale
* motor function of the hand and upper limb according to the Fugl-Meyer Motor Assessment Scale for Upper Extremity

ELIGIBILITY:
Inclusion Criteria:

* informed, voluntary consent of the patient
* age 45-80 years
* elementary (basic) gripping ability
* degree of paresis of the upper limb and hand 4 -5 on the Brunnström scale
* degree of disability on the Rankin scale 3
* spastic tension of the upper limb, paresis hand not more than 3 on the modified Ashworth scale - current health condition confirmed by a medical examination, allowing participation in tests and exercises

Exclusion Criteria:

* lack of informed, voluntary consent of the patient
* second or subsequent stroke, hemorrhagic stroke, stroke of the brainstem and cerebellum
* disorders of higher mental functions limiting comprehension and carrying out tasks during exercises
* visual field disturbances
* mechanical and thermal injuries that may limit the grasping function of the hand
* concomitant neurological, rheumatological and orthopedic diseases, including permanent - contractures that may affect the grasping ability and locomotion
* unstable medical condition
* failure to complete a 3-week rehabilitation stay

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01-19 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Motor capacities of the upper limb, according to Fugl-Meyer Motor Assessment Scale | First examination - before the start of the rehabilitation program
  It consists of 33 items assessing motor function and reflexes. The patient can score a maximum of 66 points, where each item on the scale is rated as: 0=unable, 1=partially able, or 2=fully able to perform the movement
Motor capacities of the upper limb, according to Fugl-Meyer Motor Assessment Scale | Second examination - at the end of the three-week program
  It consists of 33 items assessing motor function and reflexes. The patient can score a maximum of 66 points, where each item on the scale is rated as: 0=unable, 1=partially able, or 2=fully able to perform the movement
Motor capacities of the upper limb, according to Fugl-Meyer Motor Assessment Scale | Third study (flow-up) - 3 months after hospital discharge, during a follow-up visit
  It consists of 33 items assessing motor function and reflexes. The patient can score a maximum of 66 points, where each item on the scale is rated as: 0=unable, 1=partially able, or 2=fully able to perform the movement

SECONDARY OUTCOMES:
Hand grip strength | First examination - before the start of the rehabilitation program
  measurements to be performed with a dynamometer The dynamometer registers strength lower than up to 90 kg,
Hand grip strength | Second examination - at the end of the three-week program
  measurements to be performed with a dynamometer The dynamometer registers strength
Hand grip strength | Third study (flow-up) - 3 months after hospital discharge, during a follow-up visit
  measurements to be performed with a dynamometer The dynamometer registers strength lower than up to 90 kg,
Assessment of functional status was assessed using the Barthel Index. The subjects could score the maximum of 100 points. | First examination - before the start of the rehabilitation program
  Activities of daily living were assessed using Barthel Index. The subjects could score the maximum of 100 points.
  A maximum of 100 points can be obtained on the Barthel scale. There are three assessment ranges: getting from 0 to 20 points. means total dependence, from 20 to 80 points. means that to some extent the patient needs help from others, and the assessment in the border is 80 to 100 points. means that with a little help the patient can function alone.
  0-20 points patient's condition "light" 21-85 points - "medium-heavy" patient condition 86-100 points - patient condition "very heavy"
Assessment of functional status was assessed using the Barthel Index. The subjects could score the maximum of 100 points. | Second examination - at the end of the three-week program
  Activities of daily living were assessed using Barthel Index. The subjects could score the maximum of 100 points.
  A maximum of 100 points can be obtained on the Barthel scale. There are three assessment ranges: getting from 0 to 20 points. means total dependence, from 20 to 80 points. means that to some extent the patient needs help from others, and the assessment in the border is 80 to 100 points. means that with a little help the patient can function alone.
  0-20 points patient's condition "light" 21-85 points - "medium-heavy" patient condition 86-100 points - patient condition "very heavy"
Assessment of functional status was assessed using the Barthel Index. The subjects could score the maximum of 100 points. | Third study (flow-up) - 3 months after hospital discharge, during a follow-up visit
  Activities of daily living were assessed using Barthel Index. The subjects could score the maximum of 100 points.
  A maximum of 100 points can be obtained on the Barthel scale. There are three assessment ranges: getting from 0 to 20 points. means total dependence, from 20 to 80 points. means that to some extent the patient needs help from others, and the assessment in the border is 80 to 100 points. means that with a little help the patient can function alone.
  0-20 points patient's condition "light" 21-85 points - "medium-heavy" patient condition 86-100 points - patient condition "very heavy"
Manual skills, assessed with Box and Blocks test; | First examination - before the start of the rehabilitation program
  The test uses a wooden box, divided into two equal parts by a partition, as well as 150 blocks. The subject moves as many blocks as possible from one part of the box to the other during 60 seconds.
Manual skills, assessed with Box and Blocks test; | Second examination - at the end of the three-week program
  The test uses a wooden box, divided into two equal parts by a partition, as well as 150 blocks. The subject moves as many blocks as possible from one part of the box to the other during 60 seconds.
Manual skills, assessed with Box and Blocks test; | Third study (flow-up) - 3 months after hospital discharge, during a follow-up visit
  The test uses a wooden box, divided into two equal parts by a partition, as well as 150 blocks. The subject moves as many blocks as possible from one part of the box to the other during 60 seconds.
Assessment of proprioception Thumb Localizing Test (TLT) | First examination - before the start of the rehabilitation program
  . Thumb Localizing Test (TLT). (A) positioning of the paretic UE by the examiner. (B) four spaces in which the paretic UE is placed. Distal spaces are not far from the trunk because the reaching limb should be able to reach them without difficulty. (C) rating of positive results.
Assessment of proprioception Thumb Localizing Test (TLT) | Second examination - at the end of the three-week program
  . Thumb Localizing Test (TLT). (A) positioning of the paretic UE by the examiner. (B) four spaces in which the paretic UE is placed. Distal spaces are not far from the trunk because the reaching limb should be able to reach them without difficulty. (C) rating of positive results.
Assessment of proprioception Thumb Localizing Test (TLT) | Third study (flow-up) - 3 months after hospital discharge, during a follow-up visit
  . Thumb Localizing Test (TLT). (A) positioning of the paretic UE by the examiner. (B) four spaces in which the paretic UE is placed. Distal spaces are not far from the trunk because the reaching limb should be able to reach them without difficulty. (C) rating of positive results.
Proprioception was assessed using a mirror tester for elbow flexion and dorsal and palmar flexion of the radiocarpal joint | First examination - before the start of the rehabilitation program
  Assessments were performed with eyes closed. Proprioception of the elbow joint was assessed in the 60° elbow flexion position using a plastic Jamar goniometer. The initial fixed axis of the goniometer was set at the lateral epicondyle of the humerus, and the mobile axis was set parallel to the radius, in accordance with the methodology of the study of joint position sensation in the elbow
Proprioception was assessed using a mirror tester for elbow flexion and dorsal and palmar flexion of the radiocarpal joint | Second examination - at the end of the three-week program
  Assessments were performed with eyes closed. Proprioception of the elbow joint was assessed in the 60° elbow flexion position using a plastic Jamar goniometer. The initial fixed axis of the goniometer was set at the lateral epicondyle of the humerus, and the mobile axis was set parallel to the radius, in accordance with the methodology of the study of joint position sensation in the elbow
Proprioception was assessed using a mirror tester for elbow flexion and dorsal and palmar flexion of the radiocarpal joint | Third study (flow-up) - 3 months after hospital discharge, during a follow-up visit
  Assessments were performed with eyes closed. Proprioception of the elbow joint was assessed in the 60° elbow flexion position using a plastic Jamar goniometer. The initial fixed axis of the goniometer was set at the lateral epicondyle of the humerus, and the mobile axis was set parallel to the radius, in accordance with the methodology of the study of joint position sensation in the elbow
Handgrip function, according Frenchay scale | First examination - before the start of the rehabilitation program
  The scale consists of 7 tasks (pass/fail grading); the patient is awarded 1 point for each activity performed successfully, or 0 points for a failure to perform. The maximum score of seven points may be achieved for the performance of the tasks. Higher score corresponds to better manual skills. The scale measures the proximal control of the upper limb and the manual skills.
Handgrip function, according Frenchay scale | Second examination - at the end of the three-week program
  The scale consists of 7 tasks (pass/fail grading); the patient is awarded 1 point for each activity performed successfully, or 0 points for a failure to perform. The maximum score of seven points may be achieved for the performance of the tasks. Higher score corresponds to better manual skills. The scale measures the proximal control of the upper limb and the manual skills.
Handgrip function, according Frenchay scale | Third study (flow-up) - 3 months after hospital discharge, during a follow-up visit
  The scale consists of 7 tasks (pass/fail grading); the patient is awarded 1 point for each activity performed successfully, or 0 points for a failure to perform. The maximum score of seven points may be achieved for the performance of the tasks. Higher score corresponds to better manual skills. The scale measures the proximal control of the upper limb and the manual skills.

OTHER OUTCOMES:
Assessment of muscle tone (spasticity) was examined with modified Ashworth scale. | First examination - before the start of the rehabilitation program
  Increased muscle tone (spasticity) was examined with modified Ashworth scale. This is a six-point scale modified to include grade 1.
  0: No increase in muscle tone
  Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension 1+: Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved Considerable increase in muscle tone, passive movement difficult Affected part(s) rigid in flexion or extension [Time Frame: First examination - before the start of the rehabilitation program]
Assessment of disability level, using the modified Rankin scale (MRS) | First examination - before the start of the rehabilitation program
  Assessment of disability using the modified Rankin scale (MRS)
  Score Description 0 - No symptoms at all
  1- No significant disability despite symptoms; able to carry out all usual duties and activities 2 - Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance 3 - Moderate disability; requiring some help, but able to walk without assistance 4 - Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance 5 - Severe disability; bedridden, incontinent and requiring constant nursing care and attention 6 - Dead TOTAL (0-6):
Assessment of paretic limb function was assessed using the Brunnström scale | First examination - before the start of the rehabilitation program
  Motor performance (function) of extremities was assessed using Brunnström scale. This is a six-point scale designed to assess performance (function) of paretic extremities
Body mass index (BMI) | First examination - before the start of the rehabilitation program
  WHO BMI classification for adults:
  < 18.5 - Underweight (including: <16.0 starvation, 16.0-16.9 emaciation, 17.0-18.4 underweight) 18.5-24.9 - Normal body weight 25.0-29.9 - Overweight 30.0-34.9 - Class I obesity 35.0-39.9 - Class II obesity (clinical obesity)
  ≥ 40.0 - Class III obesity (extreme obesity)

CONTACTS AND LOCATIONS:
Overall Officials: Justyna Leszczak, PhD, Principal Investigator — Univeristy of Rzeszów
Locations (1):
- University of Rzeszów, Rzeszów, Poland